CLINICAL TRIAL: NCT00624858
Title: An Open-Label Study Assessing the Safety and Efficacy of Naltrexone Sustained Release (SR)/Bupropion Sustained Release (SR) in Overweight or Obese Subjects With Major Depression
Brief Title: A Study of Naltrexone SR/ Bupropion SR in Overweight or Obese Subjects With Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB-402
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Depression
Keywords: Depression; depressed; overweight; obese
MeSH Terms: conditions — Depression; Consciousness Disorders; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NB32 (Experimental): Naltrexone SR 32 mg/Bupropion SR 360 mg/ day
  Interventions: Drug: naltrexone SR 32 mg/ bupropion SR 360 mg daily

INTERVENTIONS:
Drug: naltrexone SR 32 mg/ bupropion SR 360 mg daily — All subjects are to complete a 4 week titration period at which time subjects will be titrated up to a maintenance level of study drug. Subjects will then take the maintenance dose of study drug for an additional 20 weeks.
  During the study, subjects will receive ancillary therapy including advice on diet and exercise

SUMMARY:
The purpose of this study is to determine whether a combination of naltrexone SR and bupropion SR is safe and effective in the treatment of major depression in overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects must be 18 to 65 years of age;
* Have body mass index (BMI) greater or equal to 27 and less than or to equal 43kg/m2;
* Meet criteria for major depression
* Women of child-bearing potential, must be non-lactating and agree to use effective contraception throughout the study period and 30 days after discontinuation of study drug;
* Able to comply with all required study procedures and schedule;
* Able to speak and read English;
* Willing and able to give written informed consent

Exclusion Criteria:

* Obesity of known endocrine origin
* Serious medical condition
* History of drug or alcohol abuse or dependence
* Use of excluded concomitant medications
* History of surgical or device (e.g. gastric banding) intervention for obesity;
* History or predisposition to seizures
* Pregnant or breast-feeding women or planning to become pregnant during the study period or within 30 days of discontinuing study drug;
* Planned surgical procedure that can impact the conduct of the study;
* Use of investigational drug, device or procedure within 30 days prior to Screening;
* Participation in any previous clinical trial conducted by Orexigen Therapeutics;
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To assess the change in depressive symptoms as measured by Montgomery-Asberg Depression Rating Scale (MADRS) total score at 12 weeks | 12 Weeks

SECONDARY OUTCOMES:
To assess the percentage change from baseline in total body weight at 12 and 24 weeks. | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Derived] McElroy SL, Guerdjikova AI, Kim DD, Burns C, Harris-Collazo R, Landbloom R, Dunayevich E. Naltrexone/Bupropion combination therapy in overweight or obese patients with major depressive disorder: results of a pilot study. Prim Care Companion CNS Disord. 2013;15(3):PCC.12m01494. doi: 10.4088/PCC.12m01494. Epub 2013 Jun 20. PMID 24171147